CLINICAL TRIAL: NCT03881761
Title: Clinical Study of CD19/CD20 Bispecific Nanobody-derived CAR-T Cells in Refractroy/Relasped B Cell Lymphoma
Brief Title: CD19/20 Bispecific Nanobody-derived CAR-T Cells in B Cell Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Henan Cancer Hospital (Other Government)
Collaborators: Henan Hualong Biotechnology Company (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HenanCH CART 2-3
Record Dates: First submitted 2019-03-16; First posted 2019-03-19 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2019-01

CONDITIONS: B-Cell Lymphoma Stage I; Refractory; Relapsed
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Intervention Model Description: transfusion of CD19/CD20 bispecific CAR-T cells 24-72 hours after completion of FC regimen pretreatment
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- experimental arm (Experimental): CAR-T cell group
  Interventions: Biological: CD19/CD20 bispecific CAR-T cells

INTERVENTIONS:
Biological: CD19/CD20 bispecific CAR-T cells — collecting blood for CAR-T cells culture three days later, FC regimen (fludarabine 30mg/m2/d x 3, cyclophosphamide 600-800mg/m2/d x 2) another two days later, transfusing CD19/CD20 bispecific CAR-T cell with a dose of 1-3x106/kg

SUMMARY:
Evaluation the safety and efficacy of CD19/CD20 bispecific CAR-T cells in patients with relapsed/refractory B cell lymphoma

DETAILED DESCRIPTION:
CART cell therapy has become the treatment of choice for patients with relapsed/ refractory B cell lymphoma. Currently, CAR-T cells approved for relapsed/refractory B-cell lymphoma are mainly CAR19-T cells. Nearly half of patients who relapse after treatment with CAR19-T cells are caused by tumor cell antigen escape. Dual-target CAR-T cells targeting CD19 and CD20 may reduce the recurrence rate after treatment. This study was to evaluate the efficacy and safety of CD19/CD20 bispecific CAR-T cells in patients with relapsed/refractory B cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* expected lifetime>3 months
* CD19/CD20 positive relapsed/refractory B cell lymphoma
* KPS>70
* at least one measurable lesion according to RECIST 1.1
* enough function of hear, liver, kidney and bone marrow
* no history of severe allergies
* no other history of malignancy
* no other diseases that conflict with this regimen
* no serious mental illness
* patient or family member sign informed consent

Exclusion Criteria:

* Pregnant or lactating women
* Severe infectious or viral disease
* Active B or C viral hepatitis
* Patients who have used large amounts of glucocorticoids or other immunosuppressive agents during the last 4 weeks
* participated in other clinical studies in the last 3 months, or have been treated with other gene products
* Others not appropriate to participate in this study examined by the investigators

Ages: 17 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
occurrence of study related adverse events | one year
  safety of CAR-T cells

SECONDARY OUTCOMES:
objective response rate | three months
  proportion of patients with complete response and partial response
survival time of CAR-T cells in vivo | one year
  from the time of CAR-T cells transfusion to the first time that CAR-T cells could not be measured in vivo
progression-free survival | one year
  the enrollment to the first time that disease progression is detected

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Song, Dr., Study Chair — Henan Cancer Hospital
Locations (2):
- China (2):
  - Cancer Hospital Affiliate to Zhengzhou University & Henan Cancer Hospital, Zhengzhou, Henan
  - Henan Cancer Hospital, Zhengzhou, Henan